CLINICAL TRIAL: NCT04225221
Title: Ovarian Hormones, Reward Response, and Binge Eating in Bulimia Nervosa: An Experimental Design
Brief Title: Neurobiology of Bulimia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 19-2343; R21MH121726 (NIH)
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-06

CONDITIONS: Bulimia Nervosa
Keywords: bulimia nervosa; binge eating; eating disorder; estrogen
MeSH Terms: conditions — Bulimia Nervosa; Bulimia; Feeding and Eating Disorders | interventions — Estradiol; Progesterone; Leuprolide; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence A: estradiol followed by progesterone (Experimental): Participants are randomly assigned to treatment Sequence A: after achieving hormone suppression using Lupron, participants begin the addback period and take study medications for 8 weeks. During the 8 week period, participants will take placebo or estradiol or progesterone. Participants will not know when or for how long they are on active medication (i.e., estradiol or progesterone) or inactive (i.e., placebo) medication. When active medication is administered, participants randomized to treatment sequence A will receive estradiol addback first, followed by progesterone.
  Estradiol and progesterone are never given simultaneously. Participants are on active medication for a total of 4 weeks.
  Interventions: Drug: Estradiol; Drug: Micronized progesterone; Drug: Leuprolide Acetate; Drug: Placebo Oral Capsule
- Sequence B: progesterone followed by estradiol (Experimental): Participants are randomly assigned to treatment Sequence B: after achieving hormone suppression using Lupron, participants begin the addback period and take study medications for 8 weeks. During the 8 week period, participants will take placebo or estradiol or progesterone. Participants will not know when or for how long they are on active medication (i.e., estradiol or progesterone) or inactive (i.e., placebo) medication. When active medication is administered, participants randomized to treatment sequence B will receive progesterone first followed by estradiol.
  Estradiol and progesterone are never given simultaneously. Participants are on active medication for a total of 4 weeks.
  Interventions: Drug: Estradiol; Drug: Micronized progesterone; Drug: Leuprolide Acetate; Drug: Placebo Oral Capsule

INTERVENTIONS:
Drug: Estradiol — During estradiol administration, 2mg of estradiol is given twice daily via oral capsule.
  Other Names: E2; Estrace
Drug: Micronized progesterone — During progesterone administration, 200mg of progesterone is given twice daily via oral capsule.
  Other Names: P4; Prometrium
Drug: Leuprolide Acetate — Initial 3.75 mg intramuscular injection administered approximately Day 6 of menstrual cycle and then monthly thereafter for a total of 3 months.
  Other Names: Lupron Depot
Drug: Placebo Oral Capsule — Placebo is administered during the addback phase when participants are not taking active medication. Placebo is given so that medication administration occurs throughout the entire 8-week addback period in order to blind participants to when and for how long they are on the active medication.
  Other Names: Sugar pill

SUMMARY:
This pilot study experimentally manipulates ovarian hormones to examine the direct impact of estrogen (E2) and progesterone (P4) on binge eating symptom burden and the behavioral reward response in women with bulimia nervosa (n=15). This is completed by taking medications that change ovarian hormone levels. This line of research could lead to the development of pharmacological interventions developed to target specific areas of the brain, brain receptors, or pathways identified to be involved in the mechanism underlying ovarian hormone change and binge eating.

DETAILED DESCRIPTION:
Eating disorders (EDs) affect 15 million women in the United States and have one of the highest mortality rates of any mental illness. Despite this, the underlying neurobiology remains poorly understood. EDs predominantly occur in women, and the frequency of certain symptoms change in a predictable pattern over the menstrual cycle; specifically, symptom changes appear to be triggered by normal fluctuations in the ovarian hormones estradiol (E2) and progesterone (P4).

The objective of this study is to examine the direct and mechanistic role of E2 and P4 on binge eating in women with bulimia nervosa (BN; n = 15). The experimental design parallels an established design developed to determine the hormonal triggers of premenstrual dysphoric disorder and depression: temporarily stopping the menstrual cycle using a Gonadotropin-releasing hormone (GnRH) agonist (Lupron) and addback E2 and P4 independently in a double-blind crossover design. The overarching hypothesis is that BN represents a hormone-sensitive phenotype, and this sensitivity is modulated by E2's effects on aspects of the reward response such that reward-motivated behaviors increase in the context of low E2. This line of research will provide direction for future research addressing neuroendocrine, neurobiological, and brain activity and function in BN. To date, there are no medications that have been developed specifically for the treatment of individuals with BN.

Our specific aims are to:

Aim 1: Quantify the direct effect of E2 and P4 on binge eating in women with BN.

Aim 2: Determine the effect of E2 on reward response in women with BN.

Aim 3: Examine the association between reward response and binge eating before and after E2 addback.

ELIGIBILITY:
Inclusion Criteria

Participants will be women aged 18-42 with a current DSM-5 bulimia nervosa (BN) diagnosis who meet the below criteria. Only participants capable of giving informed consent and understanding the risks associated with the study will be enrolled.

* A regular menstrual cycle for at least three months
* < 35 BMI > 18.5
* Free of medication or medical condition that impacts ovarian hormones or is contraindicated for use with study interventions (including birth control pills)
* Speaks English

Exclusion Criteria

Patients will not be permitted to enter this protocol if they have any of the following:

* peanut allergy
* bipolar or psychotic disorder;
* current substance use disorder or frequent binge drinking behavior;
* frequent diuretic or laxative use, ipecac use;
* currently smoking > 10 cigarettes daily;
* history of a suicide attempt or current suicidal ideation;
* endometriosis;
* abnormal genital/vaginal bleeding;
* undiagnosed enlargement of the ovaries;
* liver disease;
* breast cancer;
* personal history of blood clots (a history of blood clots in the legs or lungs; DVT); pregnancy related blood clots
* history of seizures or epilepsy;
* porphyria;
* diabetes mellitus;
* malignant melanoma;
* gallbladder or pancreatic disease;
* heart or kidney disease;
* cerebrovascular disease (stroke);
* history of osteoporosis or osteopenia;
* recurrent migraine with aura;
* first degree relative (immediate family) with premenopausal breast cancer or breast cancer presenting in both breasts or any woman who has multiple family members (greater than three relatives) with postmenopausal breast cancer will also be excluded from participating in this protocol;
* Refusal to use non-hormonal contraception throughout study;
* Pregnant women will be excluded from participation (patients will be warned not to become pregnant during the study and will be advised to employ barrier contraceptive methods), and women who become pregnant (although unlikely because of the hormone manipulation) will be withdrawn;
* Any condition or symptoms considered by the study team to detrimentally impact subject safety.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Men will not be included in this study given the stated purpose of studying the impact of ovarian hormones.
Enrollment: 10 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Baker, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 18 to 24 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: SAP, Analytic Code
Time Frame: Deidentified individual data that supports the results will be shared beginning 18 to 24 months following publication.
Access Criteria: Approval from an IRB, IEC, or REB, as applicable and execution of a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Baker JH, Girdler SS, Bulik CM. The role of reproductive hormones in the development and maintenance of eating disorders. Expert Rev Obstet Gynecol. 2012 Nov 1;7(6):573-583. doi: 10.1586/eog.12.54. PMID 23585773
- [Background] Edler C, Lipson SF, Keel PK. Ovarian hormones and binge eating in bulimia nervosa. Psychol Med. 2007 Jan;37(1):131-41. doi: 10.1017/S0033291706008956. Epub 2006 Oct 12. PMID 17038206
- [Background] Klump KL, Keel PK, Culbert KM, Edler C. Ovarian hormones and binge eating: exploring associations in community samples. Psychol Med. 2008 Dec;38(12):1749-57. doi: 10.1017/S0033291708002997. Epub 2008 Feb 29. PMID 18307829
- [Background] Lester NA, Keel PK, Lipson SF. Symptom fluctuation in bulimia nervosa: relation to menstrual-cycle phase and cortisol levels. Psychol Med. 2003 Jan;33(1):51-60. doi: 10.1017/s0033291702006815. PMID 12537036
- [Background] Price WA, Torem MS, DiMarzio LR. Premenstrual exacerbation of bulimia. Psychosomatics. 1987 Jul;28(7):378-9. doi: 10.1016/s0033-3182(87)72511-0. No abstract available. PMID 3438453
- [Background] Mac Neil BA, Hudson CC, Dempsey K, Nadkarni P. A case of symptom relapse post placement of intrauterine device (IUD) in a patient with bulimia nervosa: consequence or coincidence. Eat Weight Disord. 2017 Jun;22(2):369-372. doi: 10.1007/s40519-017-0391-z. Epub 2017 Apr 24. No abstract available. PMID 28439806
- [Background] Barth C, Villringer A, Sacher J. Sex hormones affect neurotransmitters and shape the adult female brain during hormonal transition periods. Front Neurosci. 2015 Feb 20;9:37. doi: 10.3389/fnins.2015.00037. eCollection 2015. PMID 25750611
- [Background] Yoest KE, Cummings JA, Becker JB. Estradiol, dopamine and motivation. Cent Nerv Syst Agents Med Chem. 2014;14(2):83-9. doi: 10.2174/1871524914666141226103135. PMID 25540977
- [Background] Frank GK. Advances from neuroimaging studies in eating disorders. CNS Spectr. 2015 Aug;20(4):391-400. doi: 10.1017/S1092852915000012. Epub 2015 Apr 23. PMID 25902917
- [Background] Richard JE, Lopez-Ferreras L, Anderberg RH, Olandersson K, Skibicka KP. Estradiol is a critical regulator of food-reward behavior. Psychoneuroendocrinology. 2017 Apr;78:193-202. doi: 10.1016/j.psyneuen.2017.01.014. Epub 2017 Jan 28. PMID 28214679
- [Background] Klump KL, Fowler N, Mayhall L, Sisk CL, Culbert KM, Burt SA. Estrogen moderates genetic influences on binge eating during puberty: Disruption of normative processes? J Abnorm Psychol. 2018 Jul;127(5):458-470. doi: 10.1037/abn0000352. Epub 2018 Jun 21. PMID 29927265
- [Background] Schmidt PJ, Nieman LK, Danaceau MA, Adams LF, Rubinow DR. Differential behavioral effects of gonadal steroids in women with and in those without premenstrual syndrome. N Engl J Med. 1998 Jan 22;338(4):209-16. doi: 10.1056/NEJM199801223380401. PMID 9435325
- [Background] Bloch M, Schmidt PJ, Danaceau M, Murphy J, Nieman L, Rubinow DR. Effects of gonadal steroids in women with a history of postpartum depression. Am J Psychiatry. 2000 Jun;157(6):924-30. doi: 10.1176/appi.ajp.157.6.924. PMID 10831472
- [Background] Ben Dor R, Harsh VL, Fortinsky P, Koziol DE, Rubinow DR, Schmidt PJ. Effects of pharmacologically induced hypogonadism on mood and behavior in healthy young women. Am J Psychiatry. 2013 Apr;170(4):426-33. doi: 10.1176/appi.ajp.2012.12010117. PMID 23545794
- [Background] Lee EE, Nieman LK, Martinez PE, Harsh VL, Rubinow DR, Schmidt PJ. ACTH and cortisol response to Dex/CRH testing in women with and without premenstrual dysphoria during GnRH agonist-induced hypogonadism and ovarian steroid replacement. J Clin Endocrinol Metab. 2012 Jun;97(6):1887-96. doi: 10.1210/jc.2011-3451. Epub 2012 Mar 30. PMID 22466349
- [Background] Nobles CJ, Thomas JJ, Valentine SE, Gerber MW, Vaewsorn AS, Marques L. Association of premenstrual syndrome and premenstrual dysphoric disorder with bulimia nervosa and binge-eating disorder in a nationally representative epidemiological sample. Int J Eat Disord. 2016 Jul;49(7):641-50. doi: 10.1002/eat.22539. Epub 2016 May 20. PMID 27206163
- [Background] Damario MA, Hammitt DG, Galanits TM, Session DR, Dumesic DA. Pronuclear stage cryopreservation after intracytoplasmic sperm injection and conventional IVF: implications for timing of the freeze. Fertil Steril. 1999 Dec;72(6):1049-54. doi: 10.1016/s0015-0282(99)00444-6. PMID 10593380
- [Background] Bourgain C, Devroey P, Van Waesberghe L, Smitz J, Van Steirteghem AC. Effects of natural progesterone on the morphology of the endometrium in patients with primary ovarian failure. Hum Reprod. 1990 Jul;5(5):537-43. doi: 10.1093/oxfordjournals.humrep.a137138. PMID 2394784
- [Background] Berman KF, Schmidt PJ, Rubinow DR, Danaceau MA, Van Horn JD, Esposito G, Ostrem JL, Weinberger DR. Modulation of cognition-specific cortical activity by gonadal steroids: a positron-emission tomography study in women. Proc Natl Acad Sci U S A. 1997 Aug 5;94(16):8836-41. doi: 10.1073/pnas.94.16.8836. PMID 9238064
- [Background] Bloch M, Rubinow DR, Schmidt PJ, Lotsikas A, Chrousos GP, Cizza G. Cortisol response to ovine corticotropin-releasing hormone in a model of pregnancy and parturition in euthymic women with and without a history of postpartum depression. J Clin Endocrinol Metab. 2005 Feb;90(2):695-9. doi: 10.1210/jc.2004-1388. Epub 2004 Nov 16. PMID 15546899
- [Background] Roca CA, Schmidt PJ, Deuster PA, Danaceau MA, Altemus M, Putnam K, Chrousos GP, Nieman LK, Rubinow DR. Sex-related differences in stimulated hypothalamic-pituitary-adrenal axis during induced gonadal suppression. J Clin Endocrinol Metab. 2005 Jul;90(7):4224-31. doi: 10.1210/jc.2004-2525. Epub 2005 May 10. PMID 15886244
- [Background] Schmidt PJ, Steinberg EM, Negro PP, Haq N, Gibson C, Rubinow DR. Pharmacologically induced hypogonadism and sexual function in healthy young women and men. Neuropsychopharmacology. 2009 Feb;34(3):565-76. doi: 10.1038/npp.2008.24. Epub 2008 Mar 19. PMID 18354393
- [Background] Schmidt PJ, Martinez PE, Nieman LK, Koziol DE, Thompson KD, Schenkel L, Wakim PG, Rubinow DR. Premenstrual Dysphoric Disorder Symptoms Following Ovarian Suppression: Triggered by Change in Ovarian Steroid Levels But Not Continuous Stable Levels. Am J Psychiatry. 2017 Oct 1;174(10):980-989. doi: 10.1176/appi.ajp.2017.16101113. Epub 2017 Apr 21. PMID 28427285
- [Background] Naessen S, Carlstrom K, Bystrom B, Pierre Y, Hirschberg AL. Effects of an antiandrogenic oral contraceptive on appetite and eating behavior in bulimic women. Psychoneuroendocrinology. 2007 Jun;32(5):548-54. doi: 10.1016/j.psyneuen.2007.03.008. Epub 2007 May 2. PMID 17475412
- [Background] Rice VC, Richard-Davis G, Saleh AA, Ginsburg KA, Mammen EF, Moghissi K, Leach R. Fibrinolytic parameters in women undergoing ovulation induction. Am J Obstet Gynecol. 1993 Dec;169(6):1549-53. doi: 10.1016/0002-9378(93)90434-k. PMID 8267060
- [Background] Misra M, Katzman DK, Estella NM, Eddy KT, Weigel T, Goldstein MA, Miller KK, Klibanski A. Impact of physiologic estrogen replacement on anxiety symptoms, body shape perception, and eating attitudes in adolescent girls with anorexia nervosa: data from a randomized controlled trial. J Clin Psychiatry. 2013 Aug;74(8):e765-71. doi: 10.4088/JCP.13m08365. PMID 24021517
- [Background] Stampfer MJ, Colditz GA, Willett WC, Manson JE, Rosner B, Speizer FE, Hennekens CH. Postmenopausal estrogen therapy and cardiovascular disease. Ten-year follow-up from the nurses' health study. N Engl J Med. 1991 Sep 12;325(11):756-62. doi: 10.1056/NEJM199109123251102. PMID 1870648
- [Background] Lukaszuk K, Liss J, Lukaszuk M, Maj B. Optimization of estradiol supplementation during the luteal phase improves the pregnancy rate in women undergoing in vitro fertilization-embryo transfer cycles. Fertil Steril. 2005 May;83(5):1372-6. doi: 10.1016/j.fertnstert.2004.11.055. PMID 15866571
- [Background] Fatemi HM, Kolibianakis EM, Camus M, Tournaye H, Donoso P, Papanikolaou E, Devroey P. Addition of estradiol to progesterone for luteal supplementation in patients stimulated with GnRH antagonist/rFSH for IVF: a randomized controlled trial. Hum Reprod. 2006 Oct;21(10):2628-32. doi: 10.1093/humrep/del117. Epub 2006 Jul 20. PMID 16857887
- [Background] Friedler S, Raziel A, Schachter M, Strassburger D, Bukovsky I, Ron-El R. Luteal support with micronized progesterone following in-vitro fertilization using a down-regulation protocol with gonadotrophin-releasing hormone agonist: a comparative study between vaginal and oral administration. Hum Reprod. 1999 Aug;14(8):1944-8. doi: 10.1093/humrep/14.8.1944. PMID 10438404
- [Background] Humaidan P, Bredkjaer HE, Bungum L, Bungum M, Grondahl ML, Westergaard L, Andersen CY. GnRH agonist (buserelin) or hCG for ovulation induction in GnRH antagonist IVF/ICSI cycles: a prospective randomized study. Hum Reprod. 2005 May;20(5):1213-20. doi: 10.1093/humrep/deh765. Epub 2005 Mar 10. PMID 15760966
- [Background] Mitwally MF, Gotlieb L, Casper RF. Prevention of bone loss and hypoestrogenic symptoms by estrogen and interrupted progestogen add-back in long-term GnRH-agonist down-regulated patients with endometriosis and premenstrual syndrome. Menopause. 2002 Jul-Aug;9(4):236-41. doi: 10.1097/00042192-200207000-00004. PMID 12082359
- [Background] Wyatt KM, Dimmock PW, Ismail KM, Jones PW, O'Brien PM. The effectiveness of GnRHa with and without 'add-back' therapy in treating premenstrual syndrome: a meta analysis. BJOG. 2004 Jun;111(6):585-93. doi: 10.1111/j.1471-0528.2004.00135.x. PMID 15198787
- [Background] Forbush KT, Wildes JE, Pollack LO, Dunbar D, Luo J, Patterson K, Petruzzi L, Pollpeter M, Miller H, Stone A, Bright A, Watson D. Development and validation of the Eating Pathology Symptoms Inventory (EPSI). Psychol Assess. 2013 Sep;25(3):859-78. doi: 10.1037/a0032639. Epub 2013 Jul 1. PMID 23815116
- [Background] Franken IH, Muris P, Georgieva I. Gray's model of personality and addiction. Addict Behav. 2006 Mar;31(3):399-403. doi: 10.1016/j.addbeh.2005.05.022. Epub 2005 Jun 16. PMID 15964149
- [Background] Harrison A, O'Brien N, Lopez C, Treasure J. Sensitivity to reward and punishment in eating disorders. Psychiatry Res. 2010 May 15;177(1-2):1-11. doi: 10.1016/j.psychres.2009.06.010. Epub 2010 Apr 9. PMID 20381877
- [Background] Knutson B, Westdorp A, Kaiser E, Hommer D. FMRI visualization of brain activity during a monetary incentive delay task. Neuroimage. 2000 Jul;12(1):20-7. doi: 10.1006/nimg.2000.0593. PMID 10875899

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A: Estradiol Followed by Progesterone: Participants are randomly assigned to treatment Sequence A: after achieving hormone suppression using Lupron, participants begin the addback period and take study medications for 8 weeks. During the 8 week period, participants will take placebo or estradiol or progesterone. Participants will not know when or for how long they are on active medication (i.e., estradiol or progesterone) or inactive (i.e., placebo) medication. When active medication is administered, participants randomized to treatment sequence A will receive estradiol addback first, followed by progesterone.
  Estradiol and progesterone are never given simultaneously. Participants are on active medication for a total of 4 weeks.
  Estradiol: During estradiol administration, 2mg of estradiol is given twice daily via oral capsule.
  Micronized progesterone: During progesterone administration, 200mg of progesterone is given twice daily via oral capsule.
  Leuprolide Acetate: Initial 3.75 mg intramuscular injection administered approximately Day 6 of menstrual cycle and then monthly thereafter for a total of 3 months.
  Placebo Oral Capsule: Placebo is administered during the addback phase when participants are not taking active medication. Placebo is given so that medication administration occurs throughout the entire 8-week addback period in order to blind participants to when and for how long they are on the active medication.
- Sequence B: Progesterone Followed by Estradiol: Participants are randomly assigned to treatment Sequence B: after achieving hormone suppression using Lupron, participants begin the addback period and take study medications for 8 weeks. During the 8 week period, participants will take placebo or estradiol or progesterone. Participants will not know when or for how long they are on active medication (i.e., estradiol or progesterone) or inactive (i.e., placebo) medication. When active medication is administered, participants randomized to treatment sequence B will receive progesterone first followed by estradiol.
  Estradiol and progesterone are never given simultaneously. Participants are on active medication for a total of 4 weeks.
  Estradiol: During estradiol administration, 2mg of estradiol is given twice daily via oral capsule.
  Micronized progesterone: During progesterone administration, 200mg of progesterone is given twice daily via oral capsule.
  Leuprolide Acetate: Initial 3.75 mg intramuscular injection administered approximately Day 6 of menstrual cycle and then monthly thereafter for a total of 3 months.
  Placebo Oral Capsule: Placebo is administered during the addback phase when participants are not taking active medication. Placebo is given so that medication administration occurs throughout the entire 8-week addback period in order to blind participants to when and for how long they are on the active medication.
Period: Lupron and Placebo Baseline (6 Weeks)
Arm/Group | Sequence A: Estradiol Followed by Progesterone | Sequence B: Progesterone Followed by Estradiol
Started (One participant experienced a topical skin reaction to the Lupron injection and received only 1 Lupron injection and no placebo during the first period. The participant completed a shortened phase of Lupron alone for 2 weeks and proceeded directly to the first intervention followed by the second intervention (with no washout in between). Because this participant did not complete the full 6-weeks, they are counted as not complete.) | 6 | 4
Completed | 5 | 4
Not Completed | 1 | 0
Period: First Intervention (2 Weeks)
Arm/Group | Sequence A: Estradiol Followed by Progesterone | Sequence B: Progesterone Followed by Estradiol
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Sequence A: Estradiol Followed by Progesterone | Sequence B: Progesterone Followed by Estradiol
Started (One participant experienced a topical skin reaction to the Lupron injection and received only 1 Lupron injection. The participant remained on Lupron alone for 2 weeks and proceeded directly to the first intervention followed by the second intervention (with no washout in between).) | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Sequence A: Estradiol Followed by Progesterone | Sequence B: Progesterone Followed by Estradiol
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A: Estradiol Followed by Progesterone | Sequence B: Progesterone Followed by Estradiol | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26 (7.5) | 20 (1.6) | 24 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 2 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Binge Eating Sum Score
Description: Binge eating will be measured using the 8-item binge eating subscale of the Eating Pathology Symptoms Inventory (EPSI), which measures features of binge eating (e.g., consumption of large quantities of food, mindless eating) on a 5-point Likert scale from "never" to "very often." The EPSI scale is designed to assess behavior over the past 28 days; however, to be sensitive to the timeframe of the present study, the instructions will be modified to ask participants to consider the past week. Items are summed for a scale score ranging from 0-32. Higher scores indicate more frequent experiences with binge eating behavior. Change is defined by an average change score.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of each intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Estradiol: Participants are randomly assigned to treatment Sequence A: after achieving hormone suppression using Lupron, participants begin the addback period and take study medications for 8 weeks. During the 8 week period, participants will take placebo or estradiol or progesterone. Participants will not know when or for how long they are on active medication (i.e., estradiol or progesterone) or inactive (i.e., placebo) medication. When active medication is administered, participants randomized to treatment sequence A will receive estradiol addback first, followed by progesterone.
  Estradiol and progesterone are never given simultaneously. Participants are on active medication for a total of 4 weeks.
  Estradiol: During estradiol administration, 2mg of estradiol is given twice daily via oral capsule.
  Micronized progesterone: During progesterone administration, 200mg of progesterone is given twice daily via oral capsule.
  Leuprolide Acetate: Initial 3.75 mg intramuscular injection administered approximately Day 6 of menstrual cycle and then monthly thereafter for a total of 3 months.
  Placebo Oral Capsule: Placebo is administered during the addback phase when participants are not taking active medication. Placebo is given so that medication administration occurs throughout the entire 8-week addback period in order to blind participants to when and for how long they are on the active medication.
- Progesterone: Participants are randomly assigned to treatment Sequence B: after achieving hormone suppression using Lupron, participants begin the addback period and take study medications for 8 weeks. During the 8 week period, participants will take placebo or estradiol or progesterone. Participants will not know when or for how long they are on active medication (i.e., estradiol or progesterone) or inactive (i.e., placebo) medication. When active medication is administered, participants randomized to treatment sequence B will receive progesterone first followed by estradiol.
  Estradiol and progesterone are never given simultaneously. Participants are on active medication for a total of 4 weeks.
  Estradiol: During estradiol administration, 2mg of estradiol is given twice daily via oral capsule.
  Micronized progesterone: During progesterone administration, 200mg of progesterone is given twice daily via oral capsule.
  Leuprolide Acetate: Initial 3.75 mg intramuscular injection administered approximately Day 6 of menstrual cycle and then monthly thereafter for a total of 3 months.
  Placebo Oral Capsule: Placebo is administered during the addback phase when participants are not taking active medication. Placebo is given so that medication administration occurs throughout the entire 8-week addback period in order to blind participants to when and for how long they are on the active medication.
Arm/Group | Estradiol | Progesterone
Number analyzed (Participants) | 10 | 9
score on a scale | -0.60 (4.7) | 0.89 (4.7)

2. Primary Outcome: Change in Weekly Average Binge-eating Frequency
Description: Binge eating frequency is based on a daily diary of self-reported binge eating frequency. Scores can range from 0 to infinity as they represent a self-reported frequency. Subjects self-report the number of binge eating episodes they had each day. Higher numbers indicate more frequent binge eating episodes. Average weekly frequency will be determined based on daily reported binge eating frequency. Change is defined by an average change score.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of each intervention)
Measure: Mean (Standard Deviation); unit: episodes/week
Arm/Group | Estradiol | Progesterone
Number analyzed (Participants) | 10 | 9
episodes/week | -0.48 (2.6) | 1.1 (4.7)

3. Primary Outcome: Change in Self-Reported Reward Sensitivity Subscale Score During Estradiol Manipulation
Description: Sensitivity to Punishment/Sensitivity to Reward Questionnaire will be used to measure reward sensitivity during estradiol intervention. The reward sensitivity subscale will be used, which is rated on a true/false scale with scores ranging 0-24. Higher scores indicate more sensitivity to reward. Change is defined by an average change score.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol
Number analyzed (Participants) | 10
score on a scale | -0.80 (1.9)

4. Primary Outcome: Change in Response Latency to Reward During the Monetary Incentive Delay Task During Estradiol Manipulation
Description: Time (ms) between stimulus and response will be measured during the Monetary Incentive Delay (MID) task during the win trials during the estradiol intervention. During the MID task, participants need to select the correct response during "win" and "lose" conditions by pressing a button. Higher scores indicate a longer response time to the win trials. Change is defined by an average change score.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of intervention)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Estradiol
Number analyzed (Participants) | 10
ms | -9.0 (44.0)

5. Primary Outcome: Change in Delay Discounting Parameter k Using the Monetary Choice Questionnaire With Estradiol Manipulation
Description: During the estradiol intervention, participants will be asked to make a series of hypothetical choices between small, sooner (impulsive) vs. larger, later (self controlled) hypothetical monetary outcomes. k is a hyperbolic function with larger k values indicating more valuation of a larger delayed reward and smaller values indicating preference for more immediate, smaller rewards (more impulsivity). Change is defined as the average change in k.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of intervention)
Measure: Mean (Standard Deviation); unit: k value
Arm/Group | Estradiol
Number analyzed (Participants) | 10
k value | -0.0047 (0.011)

6. Primary Outcome: Change in Self-Reported Behavioral Inhibition Score During Estradiol Manipulation
Description: This measures assesses individual disposition toward avoidance of activities during the estradiol intervention. The Behavioural Inhibition subscale of the Behavioural Inhibition Scale/Behavioral Activation Scale (BIS/BAS) assesses behavioural inhibition (BI) using participant self-reports. The minimum score on the BIS subscale is 7, maximum 28. Greater scores indicate greater behavioural inhibition. Change is defined by an average change score
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol
Number analyzed (Participants) | 10
score on a scale | 0.90 (1.8)

7. Primary Outcome: Change in Behavioral Activation Score During Estradiol Manipulation
Description: This measures assesses individual disposition toward engaging in activities during the estradiol intervention. Two BIS/BAS behavioural activation (BA) subscales will be used. The BA subscales used are Fun Seeking and Drive. Each subscale is summed to get the respective subscale scores. The minimum score on BA Fun Seeking and BA Drive are minimum 4 and maximum 16. Higher scores indicate greater behavioral activation. Change is defined by an average change score.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol
Number analyzed (Participants) | 10
score on a scale
  Fun Seeking | -0.10 (0.88)
  Drive | 0 (1.4)

8. Primary Outcome: Change in Behavioral Activation Reward Responsiveness With Estradiol Manipulation
Description: This measures assesses individual disposition toward avoiding and engaging in activities during estradiol intervention. The BIS/BAS reward responsiveness subscale will be used. The minimum score on the BA Reward Responsiveness subscale is 5, maximum 20. Higher scores indicate greater reward responsiveness. Change is defined by an average change score.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol
Number analyzed (Participants) | 10
score on a scale | 0.10 (1.2)

9. Primary Outcome: Change in Behavioral Inhibition During Estradiol Administration as Assessed Through a Behavioral Task
Description: Behavioral response inhibition will be examined during a go/no-go computerized task during the estradiol intervention. Inhibitory control is defined by the response accuracy of the go no/go trials. Percent of errors is calculated as the number of "go" responses on a "no/go" trial" divided by the total number of "no/go" trials." Fewer errors ("go" response on a "no/go" trial) indicates better inhibitory control. Change is defined by an average change score.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of intervention)
Population: Data unavailable as task was not completed by one participant.
Measure: Mean (Standard Deviation); unit: percentage of errors
Arm/Group | Estradiol
Number analyzed (Participants) | 9
percentage of errors | -0.094 (0.33)

10. Primary Outcome: Correlation Between Change in Reward Response and Change in Binge Eating Before and During Estradiol Manipulation
Description: Pearson correlations between change in self-reported reward response and change in binge eating between baseline and estradiol intervention will be examined. Binge eating is defined as the sum score from the Eating Pathology Symptom Inventory (EPSI). Self-reported reward response is defined as the BAS reward responsiveness subscale score and the Sensitivity to Reward/Sensitivity to Punishment Questionnaire (SPSRQ) sensitivity to reward subscale score. Change in binge eating and change in reward response between baseline and estradiol intervention was calculated and a correlation conducted between change scores.
Time Frame: Baseline (Day 14 of baseline) to End of Intervention (Day 14 of intervention)
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | Estradiol
Number analyzed (Participants) | 10
Pearson correlation coefficient
  BAS Reward Responsiveness | -0.146
  Sensitivity to Reward | -0.132

ADVERSE EVENTS:
Time Frame: Adverse event data was tracked once participants' began receiving the Lupron and Placebo during the initial hormone suppression stage and continued through study completion (approximately 12 weeks).
Description: All unresolved adverse events were tracked by the investigator until the events were resolved, the subject was lost to follow-up, or the adverse event was otherwise explained.
Groups:
- Lupron and Placebo: Prior to receiving hormone treatment, hormone suppression is achieved using Lupron and placebo.
  Leuprolide Acetate: Initial 3.75 mg intramuscular injection administered approximately Day 6 of menstrual cycle and then monthly thereafter for a total of 3 months.
  Placebo Oral Capsule: Placebo is administered during the addback phase when participants are not taking active medication. Placebo is given so that medication administration occurs throughout the entire 8-week addback period in order to blind participants to when and for how long they are on the active medication.
Arm/Group | Estradiol | Progesterone | Lupron and Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 5/10 | 7/9 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estradiol (N=10) | Progesterone (N=9) | Lupron and Placebo (N=10)
Localized rash at injection site (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 4 (7)
Appetite increase (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Joint discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spotting (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 5 (8)
Abdominal Cramps (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (5) — Menstrual-type cramps
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hot Flashes (Endocrine disorders) | 3 (18) | 4 (10) | 6 (54)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1)
Decreased Energy Level (General disorders) | 1 (1) | 0 (0) | 0 (0)
Breast Tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (General disorders) | 0 (0) | 0 (0) | 1 (3)
Lethargic (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 0 (0) | 2 (2) | 0 (0)
Menstrual Bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 1 (1) — Felt feverish although afebrile
Temperature Dysregulation (General disorders) | 0 (0) | 1 (1) | 0 (0) — Alternating between feeling hot and cold

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, this trial was unable to enroll the number of participants needed to complete the study leading to only a very small number of participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04225221/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT04225221/ICF_001.pdf